CLINICAL TRIAL: NCT01764581
Title: Randomized Controlled Interventional Trial of Immunosuppression Modification Based on the Cylex™ ImmuKnow® Assay in Adult Liver Transplant Recipients
Brief Title: Randomized Controlled Trial of ImmuKnow in Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Matteo Ravaioli, PhD, MD, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BolognaCylex01
Record Dates: First submitted 2013-01-02; First posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2010-10

CONDITIONS: Liver Disease
Keywords: immune monitoring; immune cell function ImmuKnow; randomized controlled trial; immunosuppression management; infection; rejection; liver transplantation; Cylex
MeSH Terms: conditions — Liver Diseases; Infections; Rejection, Psychology | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus dose regulation (Experimental): Tacrolimus dose was reduced by 25% when ImmuKnow values were below 130 ng/mL ATP and increased by 25% when ImmuKnow values exceeded 450 ng/mL.
  Interventions: Procedure: Tacrolimus regulation according to ImmuKnow values
- Control (No Intervention): immunosuppressive therapy is managed either by standard practice at our center (Control)

INTERVENTIONS:
Procedure: Tacrolimus regulation according to ImmuKnow values — Tacrolimus dose was reduced by 25% when ImmuKnow values were below 130 ng/mL ATP and increased by 25% when ImmuKnow values exceeded 450 ng/mL. Further reductions or increases were made after serial measures until ImmuKnow values stabilized between 130 and 450 ng/mL ATP. The values of 130 and 450 ng/mL ATP were previously documented as thresholds for risks of infection and rejection, respectively with a value of 280 ng/mL corresponding with the greatest negative predictive value for either event
  Other Names: Prograf
  Arms: Tacrolimus dose regulation

SUMMARY:
ImmuKnow detects cell-mediated immunity in solid-organ transplant recipients undergoing immunosuppressive therapy. Increasing ImmuKnow values indicate a decrease of immunosuppression and decreasing ImmuKnow values suggest an increase of immunosuppression. The test measures the amount of ATP produced in CD4+ lymphocytes as a biomarker of lymphocyte activation. This study uses the ImmuKnow assay to proactively adjust immunosuppressive therapy in adult liver transplant recipients to reduce the risk of adverse events

DETAILED DESCRIPTION:
We performed a randomized prospective interventional trial where the Interventional group had immunosuppression modified according to ImmuKnow values. Immunosuppression was decreased by 25% if ImmuKnow values were less than 130 ng/mL ATP. Similarly, immunosuppression was increased by 25% if ImmuKnow values were greater than 450 ng/mL ATP. Immunosuppression of the Control group was managed by the Standard of Care at our institution. ImmuKnow was performed before liver transplant, after surgery and at each clinic visit with the approximate schedule: day 1; weekly, weeks 1-4; week 6; week 8; monthly, months 3-6; and months 9 and 12. ImmuKnow testing was repeated within 7 days of a suspected/confirmed rejection or infection and again within 1 week of resolution.

ELIGIBILITY:
Inclusion Criteria:

* consecutive adult liver transplant recipients at our center;
* patients not entered into other studies;
* provided consent.

Exclusion Criteria:

* available follow-up;
* consent removed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Comparison of adverse events | 12 months posttransplant
  Comparison of adverse events consisting of allograft rejection, severe infections, graft loss and death between the Control and Interventional groups

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Daniele Pinna, MD, Study Director — Department of General Surgery and Transplantation; S.Orsola-Malpighi Hospital, University of Bologna

REFERENCES:
- [Derived] Ravaioli M, Neri F, Lazzarotto T, Bertuzzo VR, Di Gioia P, Stacchini G, Morelli MC, Ercolani G, Cescon M, Chiereghin A, Del Gaudio M, Cucchetti A, Pinna AD. Immunosuppression Modifications Based on an Immune Response Assay: Results of a Randomized, Controlled Trial. Transplantation. 2015 Aug;99(8):1625-32. doi: 10.1097/TP.0000000000000650. PMID 25757214